CLINICAL TRIAL: NCT03806907
Title: IodiNe Subtraction maPpIng in the Diagnosis of chRonic Pulmonary thromboEmbolic Disease (INSPIRE): An Observational Diagnostic Study
Brief Title: Iodine Subtraction Mapping in the Diagnosis of Chronic Pulmonary Thromboembolic Disease
Acronym: INSPIRE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Andy J Swift, Principal Investigator and Wellcome Trust Clinical Fellow in Radiology and Consultant Cardiothoracic Radiologist, University of Sheffield
Other Study IDs: STH20623
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: INSITIGATE; Pulmonary Hypertension; Pulmonary embolism; Chronic Thromboembolism; Iodine Subtraction
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Computed tomography lung subtraction iodine mapping — Subtraction of the non-contrast CT from the contrast-enhance CTPA produces the CT-LSIM
  Other Names: CT-LSIM

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a severe but treatable disease that is commonly underdiagnosed. Computed tomography lung subtraction iodine mapping (CT-LSIM) in addition to standard CT pulmonary angiography (CTPA) may improve the evaluation of suspected chronic pulmonary embolism and improve the diagnostic pick up rate. The investigators aim to recruit 100 patients suspected of having CTEPH and perform CT-LSIM scans in addition to the current gold standard test of nuclear medicine test (lung single photon emission computed tomography (SPECT) imaging) as a pilot study which will contribute to and inform the definitive trial. The diagnostic accuracy of CT-LSIM and lung SPECT will be compared. The primary outcome of the full definitive study is non-inferiority of CT-LSIM versus lung SPECT imaging.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a treatable, life-threatening disease that occurs in up to 4% of patients following acute pulmonary embolism (PE)(1). The disease is characterised by remodelling of the pulmonary arteries due to poor clearance of clot. Prognosis is very poor without treatment, and pulmonary endarterectomy (PEA) is well established as the definitive and potentially curative treatment method for CTEPH.

The European Society of Cardiology recommends ventilation/perfusion single photon emission tomography (V/Q SPECT) as the first line-screening test for patients with CTEPH. The perfusion image involves injection of 99mTc labelled macroaggregated human albumin, exposing the patient to ionizing radiation and the study acquisition time is 30-40 minutes.

Evaluation of the pulmonary arterial tree by computed tomography pulmonary angiography (CTPA) and lung perfusion is required to determine the appropriate treatment strategy in chronic thromboembolic disease (CTED). Recently, there has been much interest in the application of lung perfused blood volume images using dual-energy CT (DECT) to assess lung perfusion (2, 3). However, DECT is not widely available in hospitals across the UK and V/Q SPECT remains the reference standard. The rationale, methodology and design of the IodiNe SubtracTion mappInG in the diAgnosis of chronic pulmonary ThromboEmbolic disease (INSTIGATE) study are summarised in this paper.

Rationale of the INSTIGATE study:

Computed tomography lung subtraction iodine mapping (CT-LSIM) and accompanying software is now available in routine clinical practice (Sure subtractionTM, Toshiba Medical Systems; FDA report K130960). CT-LSIM images are created using on a non-rigid registration of a low dose unenhanced thoracic CT to a CTPA, with both examinations performed during the same sitting in less than 10 minutes total scanning time. Subtraction of the non-contrast CT from the contrast-enhance CTPA produces the CT-LSIM. CT-LSIM simultaneously provide high-spatial-resolution images of the pulmonary arterial tree and parenchymal anatomy in combination with functional examination of lung perfusion.

Magnetic resonance imaging (MRI) is an alternative approach with the advantage of the lack of ionizing radiation and can produce lung perfusion maps with good diagnostic accuracy for CTED (5). MRI is relatively limited in comparison to CT in terms of availability and the lack of ability to provide an out of hours service in some centres. Recently, it has been shown that Gadolinium is deposited in the basal ganglia, the clinical significance of the retained gadolinium in the brain, if any, remains unknown (4). Further research is ongoing.

A recent meta-analysis and systematic review, highlights the diagnostic potential of CT in both screening and for surgical and interventional operability (6).

Replacement of CT for V/Q SPECT in the setting of screening for CTED would lead to a cost saving per patient. The diagnosed incidence of CTEPH is approximately 700 cases in the UK, projected to rise to about 1000 in 2025. Estimated pick up rate of perfusion defects in patients with suspected CTED is 59% at a specialist centre (pick up rates are likely to be much lower at non-specialist centres). An estimated 1186 patients are screened at specialist centres, if these patients were screened using CT instead of SPECT, significant cost savings can be made.

In patients found to have CTED on lung SPECT, CTPA is also required to characterise the extent of pulmonary arterial clot for surgical planning, and this would be a further cost. By using CTPA with iodine subtraction mapping for screening and surgical planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected to have CTED and require a SPECT and CTPA

Exclusion Criteria:

* Less than 18 years old
* Unable to provide informed consent
* Significant renal dysfunction (GFR <30ml/min)
* History of hypersensitivity to contrast material
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient suspected to have or diagnosed with chronic thromboembolic disease and require a SPECT and CTPA
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the diagnostic performance of CT-LSIM for evaluation of pulmonary perfusion in patients with known or suspected chronic thromboembolic pulmonary hypertension (CTEPH) | 12 months
  Sensitivity and specificity

SECONDARY OUTCOMES:
Diagnostic accuracy of CT-LSIM compared with single photon emission computed tomography (SPECT) | 12 months
  Sensitivity and specificity
Diagnostic accuracy of CT-LSIM compared with CT pulmonary angiography (CTPA) | 12 months
  Sensitivity and specificity
Diagnostic accuracy of experienced and less experienced observers | 12 months
  Sensitivity and specificity
Number of alternate diagnoses made on CT-LSIM over lung SPECT imaging | 12 months
  Chi square
Radiation dose between CT-LSIM, SPECT and CTPA | 12 months
  Means

CONTACTS AND LOCATIONS:
Overall Officials: David Kiely, MD, Study Director — Sheffield Teaching Hospitals NHS Foundation Trust; Yousef Shahin, MD, Study Chair — University of Sheffield; Andy J Swift, PhD, Principal Investigator — University of Sheffield; Kavitasagary Karunasaagarar, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Hoey ET, Gopalan D, Ganesh V, Agrawal SK, Qureshi N, Tasker AD, Clements L, Screaton NJ. Dual-energy CT pulmonary angiography: a novel technique for assessing acute and chronic pulmonary thromboembolism. Clin Radiol. 2009 Apr;64(4):414-9. doi: 10.1016/j.crad.2008.11.007. Epub 2009 Jan 14. No abstract available. PMID 19264187
- [Background] Hoey ET, Mirsadraee S, Pepke-Zaba J, Jenkins DP, Gopalan D, Screaton NJ. Dual-energy CT angiography for assessment of regional pulmonary perfusion in patients with chronic thromboembolic pulmonary hypertension: initial experience. AJR Am J Roentgenol. 2011 Mar;196(3):524-32. doi: 10.2214/AJR.10.4842. PMID 21343493
- [Background] Gulani V, Calamante F, Shellock FG, Kanal E, Reeder SB; International Society for Magnetic Resonance in Medicine. Gadolinium deposition in the brain: summary of evidence and recommendations. Lancet Neurol. 2017 Jul;16(7):564-570. doi: 10.1016/S1474-4422(17)30158-8. Epub 2017 Jun 13. PMID 28653648
- [Background] Rajaram S, Swift AJ, Capener D, Telfer A, Davies C, Hill C, Condliffe R, Elliot C, Hurdman J, Kiely DG, Wild JM. Diagnostic accuracy of contrast-enhanced MR angiography and unenhanced proton MR imaging compared with CT pulmonary angiography in chronic thromboembolic pulmonary hypertension. Eur Radiol. 2012 Feb;22(2):310-7. doi: 10.1007/s00330-011-2252-x. Epub 2011 Sep 2. PMID 21887483
- [Background] Dong C, Zhou M, Liu D, Long X, Guo T, Kong X. Diagnostic accuracy of computed tomography for chronic thromboembolic pulmonary hypertension: a systematic review and meta-analysis. PLoS One. 2015 Apr 29;10(4):e0126985. doi: 10.1371/journal.pone.0126985. eCollection 2015. PMID 25923810